CLINICAL TRIAL: NCT07361497
Title: ROSETTA Lung-201: A Randomized, Multicenter, Open-label Phase 3 Study of Pumitamig Monotherapy Compared to Durvalumab in Participants With Unresectable Stage III NSCLC Without Progression After Platinum-based Concurrent Chemoradiation Therapy.
Brief Title: A Study to Evaluate Pumitamig Versus Durvalumab Following Concurrent Chemoradiation Therapy in Participants With Unresectable Stage III Non-small Cell Lung Cancer (NSCLC) (ROSETTA Lung-201)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA266-0001
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Pumitamig; Locally advanced; Unresectable; Stage 3 Non-small Cell Lung Cancer (NSCLC); CA2660001
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Pumitamig
- Arm B (Active Comparator)
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Pumitamig — Specified dose on specified days
  Other Names: BMS-986545
  Arms: Arm A
Drug: Durvalumab — Specified dose on specified days
  Arms: Arm B

SUMMARY:
A study to evaluate Pumitamig versus Durvalumab following concurrent chemoradiation therapy in participants with unresectable stage III Non-small Cell Lung Cancer (NSCLC)

ELIGIBILITY:
Inclusion Criteria

* Participants must have a histologically- or cytologically-confirmed diagnoses of non-small cell lung cancer (NSCLC) with unresectable Stage III disease.
* Participants must have received at least 2 cycles of platinum-based concurrent chemotherapy (a total dose of radiation of at least 54 Gy).
* Participants must have no progressive disease (PD) following treatment with concurrent chemoradiotherapy (CCRT).
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1.

Exclusion Criteria

* Participants with non-squamous histology must not have documented Epidermal Growth Factor Receptor (EGFR) and anaplastic lymphoma kinase (ALK) rearrangements.
* Participants must not have an active autoimmune disease.
* Participants must not have significant cardiovascular impairment such as uncontrolled hypertension (despite optimal medical treatment), congestive heart failure, active coronary disease (within 6 months prior to randomization), ventricular arrhythmias, major thrombotic or embolic events or major hemorrhagic events within 6 months prior to randomization, or significant risk of pulmonary hemorrhage.
* Participants must not have advanced/clinically significant lung disease (within 6 months prior to randomization) or history of interstitial lung disease (ILD) or pneumonitis requiring treatment with systemic steroids (≥ Grade 2), or current or suspected ILD or pneumonitis.
* Participants must not have any prior anticancer therapy (outside of CCRT) for locally advanced Stage III disease.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2026-04-09 (Estimated); Primary Completion 2030-09-18 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) by blinded independent central review (BICR) (per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1) | Up to 3 years

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 9 years
PFS by investigator (per RECIST v1.1) | Up to 3 years
Objective response (OR) by BICR (per RECIST v1.1) | Up to 3 years
Disease control rate (DCR) by BICR (per RECIST v1.1) | Up to 3 years
Duration of response (DOR) by BICR (per RECIST v1.1) | Up to 3 years
Time to Response (TTR) by BICR (per RECIST v1.1) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (249):
- United States (36):
  - Local Institution - 0898, Mobile, Alabama
  - Local Institution - 0585, Golden, Colorado
  - Local Institution - 0896, Newark, Delaware
  - Local Institution - 0614, Jacksonville, Florida
  - Local Institution - 0711, Ocala, Florida
  - Local Institution - 0429, Tampa, Florida
  - Local Institution - 0756, Marietta, Georgia
  - Local Institution - 0398, Chicago, Illinois
  - Local Institution - 0850, Evanston, Illinois
  - Local Institution - 0317, Fort Wayne, Indiana
  - Local Institution - 0656, Lexington, Kentucky
  - Local Institution - 0603, Boston, Massachusetts
  - Local Institution - 0419, Flint, Michigan
  - Local Institution - 0322, Maple Grove, Minnesota
  - Local Institution - 0142, Saint Paul, Minnesota
  - Local Institution - 0900, Columbia, Missouri
  - Local Institution - 0573, Buffalo, New York
  - Local Institution - 0606, New York, New York
  - Local Institution - 0339, Westbury, New York
  - Local Institution - 0909, Westbury, New York
  - Local Institution - 0412, Cincinnati, Ohio
  - Local Institution - 0359, Cleveland, Ohio
  - Local Institution - 0597, Cleveland, Ohio
  - Local Institution - 0895, Eugene, Oregon
  - Local Institution - 0240, Nashville, Tennessee
  - Local Institution - 0480, Nashville, Tennessee
  - Local Institution - 0908, Amarillo, Texas
  - Local Institution - 0857, Austin, Texas
  - Local Institution - 0894, Denton, Texas
  - Local Institution - 0811, Fort Worth, Texas
  - Local Institution - 0596, Houston, Texas
  - Local Institution - 0902, San Antonio, Texas
  - Local Institution - 0899, Tyler, Texas
  - Local Institution - 0133, Christiansburg, Virginia
  - Local Institution - 0250, Norfolk, Virginia
  - Local Institution - 0302, Vancouver, Washington
- Argentina (8):
  - Local Institution - 0093, Buenas Aires, Buenos Aires
  - Local Institution - 0082, Mar del Plata, Buenos Aires
  - Local Institution - 0097, Rosario, Santa Fe Province
  - Local Institution - 0094, Buenos Aires
  - Local Institution - 0078, Buenos Aires
  - Local Institution - 0761, Buenos Aires
  - Local Institution - 0608, Córdoba
  - Local Institution - 0313, Córdoba
- Australia (7):
  - Local Institution - 0456, Gosford, New South Wales
  - Local Institution - 0448, Elizabeth Vale, South Australia
  - Local Institution - 0442, Ballarat, Victoria
  - Local Institution - 0458, Epping, Victoria
  - Local Institution - 0476, Joondalup, Western Australia
  - Local Institution - 0446, Kingswood, NSW
  - Local Institution - 0451, Wentworthville
- Austria (3):
  - Local Institution - 0190, Innsbruck
  - Local Institution - 0192, Linz
  - Local Institution - 0207, Vienna
- Belgium (7):
  - Local Institution - 0906, Brasschaat, Antwerpen
  - Local Institution - 0111, Gilly, Hainaut
  - Local Institution - 0714, Genk, Limburg
  - Local Institution - 0117, Sint-Niklaas, Oost-Vlaanderen
  - Local Institution - 0122, Brussels
  - Local Institution - 0120, Ghent
  - Local Institution - 0116, Leuven
- Brazil (6):
  - Local Institution - 0615, Teresina, Piauí
  - Local Institution - 0498, Natal/RN, Rio Grande do Norte
  - Local Institution - 0619, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0535, Barretos, São Paulo
  - Local Institution - 0538, São José do Rio Preto, São Paulo
  - Local Institution - 0912, São Paulo
- Bulgaria (5):
  - Local Institution - 0736, Haskovo
  - Local Institution - 0551, Rousse
  - Local Institution - 0826, Sofia
  - Local Institution - 0732, Sofia
  - Local Institution - 0838, Sofia
- Canada (3):
  - Local Institution - 0337, Ottawa, Ontario
  - Local Institution - 0644, Montreal, Quebec
  - Local Institution - 0682, Québec
- Chile (6):
  - Local Institution - 0910, Antofagasta, AN
  - Local Institution - 0855, Las Condes, Arica y Parinacota Region
  - Local Institution - 0328, Viña del Mar, Región de Valparaíso
  - Local Institution - 0478, Santiago, Santiago Metropolitan
  - Local Institution - 0037, Santiago, Santiago Metropolitan
  - Local Institution - 0077, Santiago, Santiago Metropolitan
- China (23):
  - Local Institution - 0754, Beijing, Beijing Municipality
  - Local Institution - 0308, Chongqing, Chongqing Municipality
  - Local Institution - 0245, Fuzhou, Fujian
  - Local Institution - 0298, Shantou, Guangdong
  - Local Institution - 0249, Zhengzhou, Henan
  - Local Institution - 0911, Jingzhou, Hubei
  - Local Institution - 0813, Wuhan, Hubei
  - Local Institution - 0489, Changsha, Hunan
  - Local Institution - 0254, Nanchang, Jiangxi
  - Local Institution - 0242, Shenyang, Liaoning
  - Local Institution - 0527, Xi'an, Shaanxi
  - Local Institution - 0528, Jinan, Shandong
  - Local Institution - 0297, Jinan, Shandong
  - Local Institution - 0248, Shanghai, Shanghai Municipality
  - Local Institution - 0542, Taiyuan, Shanxi
  - Local Institution - 0440, Chengdu, Sichuan
  - Local Institution - 0835, Chengdu, Sichuan
  - Local Institution - 0719, Hangzhou, Zhejiang
  - Local Institution - 0253, Linhai, Zhejiang
  - Local Institution - 0561, Guangzhou
  - Local Institution - 0301, Hangzhou
  - Local Institution - 0537, Shanghai Shi
  - Local Institution - 0564, Xi'an
- France (12):
  - Local Institution - 0023, Toulouse, Midi-Pyrénées
  - Local Institution - 0716, Lille, Nord
  - Local Institution - 0024, Amiens
  - Local Institution - 0029, Borddeaux Cedex
  - Local Institution - 0129, Dijon
  - Local Institution - 0025, Limoges
  - Local Institution - 0130, Lyon
  - Local Institution - 0028, Montpellier
  - Local Institution - 0127, Nantes
  - Local Institution - 0026, Paris
  - Local Institution - 0689, Villejuif
  - Local Institution - 0021, Paris, Île-de-France Region
- Germany (13):
  - Local Institution - 0739, Augsburg, Bavaria
  - Local Institution - 0265, Koblenz, Rhineland-Palatinate
  - Local Institution - 0174, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Local Institution - 0172, Kiel, Schleswig-Holstein
  - Local Institution - 0182, Jena, Thuringia
  - Local Institution - 0217, Berlin
  - Local Institution - 0215, Berlin
  - Local Institution - 0169, Göttingen
  - Local Institution - 0178, Gröbenzell
  - Local Institution - 0199, Haile
  - Local Institution - 0299, Hamburg
  - Local Institution - 0186, Immenhausen
  - Local Institution - 0187, Regensburg
- Greece (6):
  - Local Institution - 0416, Thessaloniki, Thessaloníki
  - Local Institution - 0321, Larissa, Thessalía
  - Local Institution - 0391, Athens
  - Local Institution - 0323, Athens
  - Local Institution - 0324, Athens
  - Local Institution - 0697, Thessaloniki
- Hong Kong (3):
  - Local Institution - 0457, Tuenmen, NT
  - Local Institution - 0193, Hksar
  - Local Institution - 0764, Shatin
- Hungary (5):
  - Local Institution - 0139, Kecskemét, Bács-Kiskun county
  - Local Institution - 0787, Szolnok, Jász-Nagykun-Szolnok
  - Local Institution - 0138, Budapest
  - Local Institution - 0776, Farkasgyepű
  - Local Institution - 0696, Törökbálint
- India (9):
  - Local Institution - 0840, Eluru, Andhra Pradesh
  - Local Institution - 0548, Pūlakkōd, Kerala
  - Local Institution - 0864, Aurangabad, Maharashtra
  - Local Institution - 0660, Mumbai, Maharashtra
  - Local Institution - 0663, Mumbai, Maharashtra
  - Local Institution - 0661, Nagpur, Maharashtra
  - Local Institution - 0657, Hyderabad, Telangana
  - Local Institution - 0547, Delhi
  - Local Institution - 0659, Pune
- Ireland (3):
  - Local Institution - 0276, Cork
  - Local Institution - 0270, Dublin
  - Local Institution - 0070, Dublin
- Italy (8):
  - Local Institution - 0304, Orbassano, Piedmont
  - Local Institution - 0669, Rome, Roma
  - Local Institution - 0269, Aviano (PN)
  - Local Institution - 0668, Milan
  - Local Institution - 0667, Milan
  - Local Institution - 0275, Napoli
  - Local Institution - 0390, Parma
  - Local Institution - 0670, Ravenna
- Japan (14):
  - Local Institution - 0014, Nagoya, Aichi-ken
  - Local Institution - 0701, Kobe, Hyōgo
  - Local Institution - 0154, Nishinomiya-shi, Hyōgo
  - Local Institution - 0001, Sendai, Miyagi
  - Local Institution - 0907, Okayama, Okayama-ken
  - Local Institution - 0002, Osakasayama-shi, Osaka
  - Local Institution - 0149, Hidaka, Saitama-Pref
  - Local Institution - 0018, Bunkyo-ku, Tokyo
  - Local Institution - 0158, Hamamatsu
  - Local Institution - 0016, Hirakata-shi
  - Local Institution - 0009, Minami-Ku, Fukuoka
  - Local Institution - 0157, Sagamihara
  - Local Institution - 0759, Sendai
  - Local Institution - 0008, Yokohama
- Mexico (6):
  - Local Institution - 0772, Saltillo, Coahuila
  - Local Institution - 0815, Tijuana, Estado de Baja California
  - Local Institution - 0699, Zapopan, Jalisco
  - Local Institution - 0330, Monterrey, Nuevo León
  - Local Institution - 0914, Puebla City
  - Local Institution - 0349, Querétaro
- Netherlands (6):
  - Local Institution - 0095, Breda, North Brabant
  - Local Institution - 0091, Amsterdam, North Holland
  - Local Institution - 0089, Groningen
  - Local Institution - 0243, Nijmegen
  - Local Institution - 0092, Tilburg
  - Local Institution - 0087, Zwolle
- Poland (4):
  - Local Institution - 0473, Lublin, Lublin Voivodeship
  - Local Institution - 0556, Przemyśl, Podkarpackie Voivodeship
  - Local Institution - 0681, Katowice, Silesian Voivodeship
  - Local Institution - 0680, Opole
- Local Institution - 0897, Peru, Puerto Rico
- Romania (7):
  - Local Institution - 0219, Bucharest, București
  - Local Institution - 0046, Bucharest
  - Local Institution - 0168, Cluj-Napoca
  - Local Institution - 0045, Craiova
  - Local Institution - 0058, Floresti/ Cluj
  - Local Institution - 0184, Iași
  - Local Institution - 0164, Iași
- Singapore (2):
  - Local Institution - 0650, Singapore, Central Singapore
  - Local Institution - 0647, Singapore
- South Korea (6):
  - Local Institution - 0151, Seongnam, Kyǒnggi-do
  - Local Institution - 0055, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0035, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0064, Seoul, Seoul-teukbyeolsi
  - Local Institution - 0052, Cheongju-si
  - Local Institution - 0063, Seoul
- Spain (9):
  - Local Institution - 0041, L'Hospitalet Del Llobregat, Barcelona [Barcelona]
  - Local Institution - 0086, Barakaldo
  - Local Institution - 0043, Barcelona
  - Local Institution - 0042, Barcelona
  - Local Institution - 0049, Madrid
  - Local Institution - 0570, Málaga
  - Local Institution - 0061, Seville
  - Local Institution - 0066, Valencia
  - Local Institution - 0044, Zaragoza
- Sweden (3):
  - Local Institution - 0033, Gävle, Gävleborgs Län [se-21]
  - Local Institution - 0032, Solna, Stockholms Län [se-01]
  - Local Institution - 0034, Uppsala
- Switzerland (3):
  - Local Institution - 0222, Basel
  - Local Institution - 0738, Münsterlingen
  - Local Institution - 0165, Sankt Gallen
- Taiwan (4):
  - Local Institution - 0735, Chiayi City
  - Local Institution - 0726, Taipei
  - Local Institution - 0734, Taipei
  - Local Institution - 0729, Taipei
- Thailand (3):
  - Local Institution - 0733, Bangkok
  - Local Institution - 0160, Khon Kaen
  - Local Institution - 0728, Songkhla
- Turkey (Türkiye) (6):
  - Local Institution - 0099, Adana
  - Local Institution - 0113, Adana
  - Local Institution - 0198, Antalya
  - Local Institution - 0109, Çankaya
  - Local Institution - 0096, Istanbul
  - Local Institution - 0107, Istanbul
- United Kingdom (11):
  - Local Institution - 0239, Manchester, Lancashire
  - Local Institution - 0672, Cambridge
  - Local Institution - 0289, Cardiff
  - Local Institution - 0557, Gloucester
  - Local Institution - 0257, Guildford
  - Local Institution - 0693, Leeds
  - Local Institution - 0232, Liverpool
  - Local Institution - 0296, London
  - Local Institution - 0235, London
  - Local Institution - 0533, Middlesex
  - Local Institution - 0913, Sutton
- Local Institution - 0856

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07361497.html